CLINICAL TRIAL: NCT07017192
Title: OPPOSED (anteriOr hiP arthroPlasty regiOnal aneSthEsia stuDy) Study. Regional Anesthesia Techniques for Anterior Approach Hip Arthroplasty Analgesia: SIFI Block Versus Lumbar ESP Block
Brief Title: OPPOSED (anteriOr hiP arthroPlasty regiOnal aneSthEsia stuDy) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77/2025
Record Dates: First submitted 2025-05-22; First posted 2025-06-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: Hip Replacement Surgery; Hip Replacement, Total; Hip Pain; Hip Arthroplasty; Hip Replacement Postoperative; Hip Surgery; Pain,Postoperative; Mobility and Independence
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects udergoing SIFI block (Experimental)
  Interventions: Procedure: SIFI Block
- Subjects udergoing ESP block (Experimental)
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: SIFI Block — Infiltration of local anesthetics in the suprainguinal iliac fascia (Ropivacaine 0.375 40 mls)
  Arms: Subjects udergoing SIFI block
Procedure: ESP block — Infiltration of local anesthetics in the fascial plane underneath the erector spoinae mulscle at lumbar level (Ropivacaine 0.375 40 mls)
  Arms: Subjects udergoing ESP block

SUMMARY:
Main indications for total hip arthroplasty (THA) are degenerative osteoarthritis of the coxofemoral joint, osteonecrosis of the hip, congenital disorders such as dysplasia and inflammatory arthritis. More recently, surgery using the direct anterior approach is getting popularity: this method, in fact, granting a significant sparing of the hip muscles, is associated with favorable results compared to other techniques, such as a lower risk of dislocation, limitated damage to soft tissues with better recovery and early discharge.

Patients undergoing this procedure may although experience moderate to severe postoperative pain in the first few hours (with peaks observed in the first 12 hours), as well as potential complications such as nausea and vomiting related to opioids use.

It has been shown that adequate pain control influences early mobilization and rehabilitation, ensuring a quicker recovery. The role of regional anesthesia techniques has been established in almost all areas of orthopedic surgery, and in particularly in the management of postoperative pain following hip replacement surgery, but definitive data are missing with regard to direct anterior approach.

Regional anesthesia consists of infiltrating local anesthetics in sites (fascial planes or nerves), in order to limit or even eliminate the use of traditional painkillers, with a significant reduction in the side effects.

The aim of this study is to compare the impact of two techniques, the Suprainguinal Fascia Iliaca (SIFI) block and the lumbar Erector Spinae Plane (ESP) block, in managing postoperative pain in subjects undergoing total hip replacement surgery performed by direct anterior approach.

The primary objective of the study is the incidence of residual femoral and obturator nerves block (knee extension and hip adduction according to ASIA score) 8 hours after surgery in the two treatment groups.

Secondary objectives include: • Time elapsed between the end of surgery and the recovery of lower limb motility enough to allow the patient to mobilize independently; • Total opioid consumption (calculated as morphine equivalents) at 8, 24 and 48 hours after surgery; • Pain according to NRS (numerica rating scale) at 8, 24 and 48 hours after surgery; • Extent of sensory block of the three branches of the lumbar plexus (femoral, obturator, lateral femorocutaneuous nerves) at 8, 24 and 48 hours after surgery; • Timing of hospital discharge; • Incidence of chronic or persistent postoperative pain (at 30 and 90 days after surgery); • Any postoperative complication

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years and =<85 years
* patients undergoing elective unilateral THA with direct anterior approach
* patients able to understand the purposes of the study and provide signed informed consent

Exclusion Criteria:

* pregnancy
* Age <18 years or >85 years
* revision or bilateral surgeries
* psychiatric pathology or cognitive deficits, mental retardation, inability to provide valid informed consent
* History of illicit drugs and/or alcohol abuse
* urgent/emergent surgery with admission to Intensive Care under sedation and mechanical ventilation or complications that do not allow evaluation
* known allergy to the drugs used in the study
* refusal to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of residual femoral and obturator nerves block in the two treatment groups | 8 hours after surgery
  (knee extension and hip adduction according to ASIA score)

SECONDARY OUTCOMES:
Time elapsed between the end of surgery and the recovery of lower limb motility | 8 (or more) hours after surgery
  Ability of patient to mobilize independently within the room
Total opioid consumption | 8, 24 and 48 hours after surgery
  Calculated as morphine equivalents
Pain according to NRS (Numeric Rating Scale) | 8, 24 and 48 hours after surgery
  Scale 1-10 (1 corresponding to minimum and 10 corresponding to maximum pain perceived)
Extent of sensory block | 8, 24 and 48 hours after surgery
  Clinical evaluation of the three branches of the lumbar plexus (femoral, obturator, lateral femorocutaneuous nerves)
Incidence of postoperative complications | Up to 48 hrs after surgery
  Bleeding, Bradyarrhythmic and/or hypotensive events, Nausea and Vomiting
Timing of hospital discharge | From enrolment to the first follow up at 30 days
Incidence of chronic or persistent postoperative pain | 30 and 90 days after surgery
  Follow-up by phone, using Brief Pain Inventory (presence of pain/localization/characteristics) and DN4 (neuropathic component) questionnaires.
Incidence of acute side effects related to opioid use | Up to 48 hours after surgery
  excessive sedation, nausea and vomiting, respiratory depression, pruritus, urinary retention, constipation
Incidence of complications related to nerve blocks | up to 48 hours after surgery
  block failure, nerve damage, hematomas, systemic toxicity from local anesthetics

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No